CLINICAL TRIAL: NCT04509960
Title: Comparison of Airway Placement Conditions and Postoperative Effects of Laryngoscope-guided Laryngeal Mask Placement Methods in Sniffing Position in Geriatric Edentulous Patients
Brief Title: Different Ways of Airway Management in Elective Minor Surgeries in Geriatric Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Diskapi Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Filiz Akaslan, specialist, Ankara Diskapi Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: LMA
Record Dates: First submitted 2020-06-13; First posted 2020-08-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Comparison of Different Laryngeal Mask Wearing Methods
Keywords: laryngeal mask

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- proseal laryngeal mask insertion (No Intervention): no intervention
- proseal laryngeal mask insertion with laryngoscope (Experimental): with the help of direct laryngoscopy
  Interventions: Device: direct laryngoskopy

INTERVENTIONS:
Device: direct laryngoskopy — Proseal Laryngeal mask inserted with direct laryngoskopy
  Arms: proseal laryngeal mask insertion with laryngoscope

SUMMARY:
different ways of airway management in elective minor surgeries of geriatric patients

DETAILED DESCRIPTION:
The investigators will used two different ways of pro-seal laryngeal mask insertion technique (laryngoscopy- guided technique or the standard technique) in elective minor surgeries of geriatric toothless patients.

The investigators will record the respiratory dynamics, heartbeat, systolic, diastolic, mean arterial pressures every 5 minutes during surgery. The investigators will record the laryngeal mask insertion time and oropharyngeal leakage pressure. The investigators will evaluate the placement of a laryngeal mask according to young criteria. The development and severity of coughing, retching, laryngospasm, extremity, and head movement during laryngeal mask placement will be recorded. Bloodstains, sore throat, hoarseness will be recorded on the mask that may develop due to laryngeal mask placement. The investigators will use the Briacombe scoring and Campbell category system to assess the position of laryngeal mask airway devices.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I or II or III
2. Who were scheduled to minor elective ambulatory surgery (e.g. urology operations)
3. Patients undergoing general anesthesia
4. Those who are planned to wear a laryngeal mask for surgical procedure

Exclusion Criteria:

1. patients with full stomach
2. A history of gastric reflux
3. A history of convulsions, cardiovascular or neuromuscular disease
4. Allergies to the study drugs
5. obese (Body mass index (BMI) ≥ 40 kg / m2)
6. suspected difficult airway and hyper-reactive airway disease

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-03-30 (Estimated); Study Completion 2021-04-30 (Estimated)

PRIMARY OUTCOMES:
laryngeal mask placement | First minute after laryngeal mask insertio
  To evaluate the best fiberoptic bronchoscopic view while insertion of pro-Seal laryngeal mask either in a classic way, or with the help of laryngoscope. The fibreoptic evaluation Includes 4, only vocal cords visible; 3, vocal cords plus posterior epiglottis visible 2, vocal cords plus anterior epiglottis visible
  ; 1, vocal cords not seen.
complications of laryngeal mask insertion | Complications will be evaluated within 1 hour after patient recovery.
  complications like sore throat, hoarseness, nausea, and vomiting or Bloodstain on the laryngeal mask.
  we simply asked patients about them

SECONDARY OUTCOMES:
hemodynamic response | Before putting on the Layngeal mask, it will record in beats / minute at 5 minutes for 1 minute and 20 minutes after wearing
  Heart rate will record before LMA and post LMA used at first minute
insertion time | The investigator will record the insertion time in seconds from the moment the laryngeal mask airway passes the incisors until the end-tidal CO2 is visible.
  Insertion time was defined from the time of removal of the facemask to the time of the appearance of first capnography upstroke. we assessed this outcome stopwatch
respiratory dynamics | The first minute after the laryngeal mask insertion, and every 5 minutes thereafter up to the 20th minute
  The investigator will record the (tidal volume(ml) value from the mechanical ventilator after wearing the laryngeal mask.
hemodynamic responce | Before putting on the Layngeal mask, it will record in mm Hg at 5 minutes for 1 minute and 20 minutes after wearing
  mean blood pressure will record before LMA and post LMA used at first minute
oxygen saturation | Before putting on the Layngeal mask, it will record in %SpO2 at 5 minutes for 1 minute and 20 minutes after wearing
  saturation will record before LMA and post LMA used at first minute
respiratory dynamics | The first minute after the laryngeal mask insertion, and every 5 minutes thereafter up to the 20th minute
  The investigator will record the peak airway pressure (cmH2O) value from the mechanical ventilator after wearing the laryngeal mask.
respiratory dynamics | The first minute after the laryngeal mask insertion, and every 5 minutes thereafter up to the 20th minute
  The investigator will record the end-tidal CO2(mmHg) value from the mechanical ventilator after wearing the laryngeal mask.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Siences Diskapi Yildirim Beyazit T&R hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandan SN, Sharma SM, Raveendra US, Rajendra Prasad B. Fiberoptic assessment of laryngeal mask airway placement: a comparison of blind insertion and insertion with the use of a laryngoscope. J Maxillofac Oral Surg. 2009 Jun;8(2):95-8. doi: 10.1007/s12663-009-0025-8. Epub 2009 Aug 11. PMID 23139483
- [Background] Kim GW, Kim JY, Kim SJ, Moon YR, Park EJ, Park SY. Conditions for laryngeal mask airway placement in terms of oropharyngeal leak pressure: a comparison between blind insertion and laryngoscope-guided insertion. BMC Anesthesiol. 2019 Jan 5;19(1):4. doi: 10.1186/s12871-018-0674-6. PMID 30611202
- [Background] Choo CY, Koay CK, Yoong CS. A randomised controlled trial comparing two insertion techniques for the Laryngeal Mask Airway Flexible in patients undergoing dental surgery. Anaesthesia. 2012 Sep;67(9):986-90. doi: 10.1111/j.1365-2044.2012.07167.x. Epub 2012 Jun 11. PMID 22686571